CLINICAL TRIAL: NCT00840853
Title: Phase I Study of the Administration of Multi-Virus-Specific Cytotoxic T Lymphocytes Expressing CD19 Chimeric Receptors for Prophylaxis or Therapy of Relapse of CD19 Positive Malignancies Post Hematopoietic Stem Cell Transplantation
Brief Title: Multi-virus CTLs Expressing CD19 Chimeric Receptors, CD19 Positive Malignancies Post SCT, MULTIPRAT
Acronym: MULTIPRAT
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Carlos Ramos, Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23637-MULTIPRAT; MultiPRAT (Other: Baylor College of Medicine)
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Acute Lymphoblastic Leukemia (ALL); Chronic Lymphocytic Leukemia (CLL); Non Hodgkin's Lymphoma
Keywords: Stem cell transplant; Acute Lymphoblastic Leukemia (ALL); Chronic Lymphocytic Leukemia (CLL); Non Hodgkin's Lymphoma; Cytotoxic T lymphocytes; CTL; CD-19; chimeric receptor
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — Diphenhydramine; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A with disease (Experimental): CD19+ B-ALL undergoing allogeneic HSCT, with minimal residual disease or relapse post-HSCT
  Patients will receive one of the following dose levels of CD19CAR/virus specific T cells:
  Dose Level 1: 1.5 x 10^7/m2
  Dose Level 2: 4.5 x 10^7/m2
  Dose Level 3: 1.2 x 10^8/m2
  Patients will be evaluated in the clinic and a single dose of CTL will be administered from day +30 post-HSCT.
  Patients may be premedicated with Benadryl and Tylenol before receiving the injection of cells.
  If patients with relapse have a partial response or have stable disease they will be eligible to receive up to 6 further doses of CTLs, each of which will consist of the same number or less than as their first injection.
  Interventions: Genetic: CD19CAR/virus specific T cells; Drug: Benadryl and Tylenol
- Group A without disease (Experimental): CD19+ B-ALL undergoing allogeneic HSCT, without detectable disease post-HSCT.
  Patients will receive CD19CAR/virus specific T cells - Dose Level 1: 1.5 x 10^7/m2
  Patients will be evaluated in the clinic and a single dose of CTL will be administered from day +30 post-HSCT.
  Patients may be premedicated with Benadryl and Tylenol before receiving the injection of cells.
  Interventions: Genetic: CD19CAR/virus specific T cells; Drug: Benadryl and Tylenol
- Group B with disease (Experimental): CD19+ B cell CLL or NHL undergoing allogeneic HSCT, with minimal residual disease or relapse post-HSCT
  Patients will receive one of the following dose levels of CD19CAR/virus specific T cells:
  Dose Level 1: 1.5 x 10^7/m2
  Dose Level 2: 4.5 x 10^7/m2
  Dose Level 3: 1.2 x 10^8/m2
  Patients will be evaluated in the clinic and a single dose of CTL will be administered from day +30 post-HSCT.
  Patients may be premedicated with Benadryl and Tylenol before receiving the injection of cells.
  If patients with relapse have a partial response or have stable disease they will be eligible to receive up to 6 further doses of CTLs, each of which will consist of the same number or less than as their first injection.
  Interventions: Genetic: CD19CAR/virus specific T cells; Drug: Benadryl and Tylenol
- Group B without disease (Experimental): CD19+ B cell CLL or NHL undergoing allogeneic HSCT, without detectable disease post-HSCT
  Patients will receive CD19CAR/virus specific T cells -
  Dose Level 1: 1.5 x 10^7/m2
  Patients will be evaluated in the clinic and a single dose of CTL will be administered from day +30 post-HSCT.
  Patients may be premedicated with Benadryl and Tylenol before receiving the injection of cells.
  Interventions: Genetic: CD19CAR/virus specific T cells; Drug: Benadryl and Tylenol

INTERVENTIONS:
Genetic: CD19CAR/virus specific T cells — CD19CAR/virus specific T cells will be thawed and given by intravenous injection from day +30 post transplant.
Drug: Benadryl and Tylenol — Patients may be premedicated with Benadryl and Tylenol before receiving the injection of cells.
  Other Names: Diphenhydramine and acetaminophen

SUMMARY:
Subjects are having a bone marrow or SCT for either a type of cancer of the blood called Leukemia or a cancer of the lymph nodes called non- Hodgkin's Lymphoma. Although a transplant can cure leukemia or lymphoma, some people will relapse. In those who relapse, current treatment cures only a very small percentage. Although giving patients a dose of donor immune cells before relapse can prevent relapse of the leukemia or lymphoma, DLI can also cause a serious complication called graft versus host disease (GVHD). This is a gene transfer research study using special immune cells which are specific for these cancer cells.

The body has different ways of fighting infection and disease. This study combines 2 of those ways, antibodies and T cells. T cells (CTLs or cytotoxic T cells) are infection-fighting blood cells that can kill cells, including tumor cells. Antibodies and T cells have been used to treat patients with cancers; they have shown promise, but haven't been strong enough to cure most patients.

The antibody used in this study is called anti-CD19. This antibody sticks to leukemia cells because of a substance on the outside of these cells called CD19. For this study, the anti-CD19 antibody has been changed so that instead of floating free in the blood it is now joined to T cells. When an antibody is joined to a T cell in this way it's called a chimeric receptor.

In the laboratory, investigators found that T cells that are trained to recognize common viruses can stay in the blood stream for many years. By joining the anti-CD19 antibody to CTLs that recognize viruses, they believe that they will also be able to make a cell that can last a long time in the body, provide protection from viruses, and recognize and kill leukemia. The CTLs which we will join the anti-CD19 antibody to attack 3 viruses (trivirus-specific CTLs), CMV, EBV, and adenovirus.

Studies have shown that trivirus-specific CTLs grown from the stem cell donor can be given safely to transplant recipients and can stop these viruses from causing severe infections. These CD19 chimeric receptor trivirus specific T cells are an investigational product not approved by the FDA.

The purpose of this study is to find the biggest dose of chimeric T cells that is safe, to assess the side effects, to see how long the T cells last and to evaluate whether this therapy might help prevent infections and relapse in people with CD19+ leukemia or lymphoma having a SCT.

DETAILED DESCRIPTION:
The donor gave us blood to make CD19 chimeric receptor trivirus specific T cells in the laboratory. These cells were grown and frozen for the subject. To make these special T cells they are grown with stimulator cells. Stimulator cells are also made from the donor's blood but they are irradiated so that they can no longer grow. Stimulator cells have been infected with viruses so that they carry proteins from 3 viruses (CMV, adenovirus, and EBV). These cells are cultured with the T cells so that they can learn to see and attack cells infected with CMV, EBV and adenovirus.

To get the CD19 antibody to attach to the surface of the T cell, an antibody gene was inserted into the T cell. This is done with a virus called a retrovirus that has been made for this study and will carry the antibody gene into the T cell. This virus also helps to find the T cells in the blood after injected. Once sufficient numbers of T cells are made, the investigators freeze the cells and test them to make sure they kill CD19+ tumors cells and cells infected with CMV, EBV and adenovirus. Once testing is completed the cells will be ready to give to the subject.

When the subject enrolls on this study, they will be assigned a dose of CD19 chimeric receptor trivirus specific T cells. The subject will be given an injection of cells into the vein through an IV line at the assigned dose. The injection will take about 20 minutes. Investigators will monitor the subject in the clinic after the injection for up to 3 hours. The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or The Methodist Hospital.

To learn more about the way the CD19 chimeric receptor trivirus specific T cells are working and how long they last in the body, extra blood will be drawn. The total blood drawn during this study will not exceed 300 tsp.

For subjects receiving the CTLs for treatment of their disease: If the subject has stable disease (the tumor did not grow) or there is a reduction in the size of the tumor on imaging studies or by blood count after the T-cell infusion, the subject can receive up to six additional doses of the T cells if they wish. After each T-cell infusion, the subject will be monitored.

Because the subject will have received cells with a new gene in them the subject will be followed for a total of 15 years to see if there are any long term side effects of gene transfer.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Any patient regardless of sex or age with CD19+ B-ALL undergoing allogeneic HSCT (Group A)

   OR Any patient regardless of sex or age with CD19+ B-CLL or NHL undergoing allogeneic HSCT (Group B).

   AND

   With minimal residual disease (MRD) or relapse post-HSCT (for the phase I dose escalation)

   OR

   With no evidence of ALL or CLL/NHL post-HSCT (to be included in the expansion cohort
2. Patients with life expectancy greater than or equal to 6 weeks
3. Patients with a Karnofsky/Lansky score greater than or equal to 50
4. Donor HIV negative
5. Patient or parent/guardian capable of providing informed consent
6. Patients with bilirubin 2x normal or less, AST 3x normal or less, creatinine less than or equal to 2x normal for age and Hgb greater than 8.0
7. Pulse oximetry of greater than 90% on room air
8. Sexually active patients must be willing to utilize one of the more effective birth control methods for 6 months after the CTL infusion. The male partner should use a condom.
9. Available allogeneic CD19CAR transduced tri-virus-specific cytotoxic T lymphocytes with greater than or equal to15% expression of CD19CAR determined by flow-cytometry and greater than 10% killing of one or more viral antigen pulsed targets in a cytotoxicity assay at an effector:target ratio of 20:1.*
10. Patients should have been off other investigational antiviral or antitumor therapy for one month prior to entry in this study.

    * Note: Cell dose is based on total cell numbers and not individual antivirus or antileukemic cell numbers.

EXCLUSION CRITERIA:

1. Severe intercurrent infection
2. Evidence of graft versus host disease >grade II
3. Pregnant or lactating
4. History of hypersensitivity reactions to murine protein-containing products.
5. Currently taking corticosteroids for therapy of GVHD.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2009-04; Primary Completion 2016-04 (Actual); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Number of dose limiting toxicities | 6 weeks
  Dose limiting toxicity (DLT) is defined as development of grade III-IV GVHD or NCI CTC grade 3-5 toxicity that is not preexisting and/or not due to the underlying malignancy or infection or treatment of relapse within 30 days of study drug administration. DLTs will be graded according to NCI CTCAE v3.0.

SECONDARY OUTCOMES:
Tumor response to gene modified CTL on measurable disease. | up to 15 years
  When appropriate, serial measurements of tumor burden will be performed either using absolute tumor cell numbers in marrow and peripheral blood or percentage of cells positive for specific cytogenetic abnormalities and/or levels of minimal residual disease by flow cytometry and molecular methods. These measures of disease activity before and after CTL infusion will be analyzed descriptively. In patients with detectable tumors and/or lymphadenopathy - response and progression will be evaluated in this study using the international criteria proposed by RECIST.
Frequency of T-cells expressing gene-modified CTLs. | up to 15 years
  To evaluate the impact of the gene modified CTL on virus-specific T-lymphocyte immune reconstitution. The repeat measurements on proliferation, immune function, etc. on each patient. Descriptive statistics using mean ± SD, medians and ranges will be calculated to summarize repeated measurements of CTL expansion, persistence, and function following infusion. Immune response to viral and leukemic antigens measured by ELISPOT will be analyzed. Plots of growth curves will be generated to graphically illustrate patterns of survival and expansion of T cells as well as immune response.
Frequency of CD19+ B-Cells post HSCT expressing gene-modified CTLs | up to 15 years
  To evaluate the impact of the gene modified CTL on normal CD19+ B-cell immune reconstitution post-HSCT. The repeat measurements on proliferation, immune function, etc. on each patient will be analyzed. Descriptive statistics using mean ± SD, medians and ranges will be calculated to summarize repeated measurements of CTL expansion, persistence, and function following infusion. Immune response to viral and leukemic antigens measured by ELISPOT will be analyzed. Plots of growth curves will be generated to graphically illustrate patterns of survival and expansion of T cells as well as immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Ramos, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Sun J, Huye LE, Lapteva N, Mamonkin M, Hiregange M, Ballard B, Dakhova O, Raghavan D, Durett AG, Perna SK, Omer B, Rollins LA, Leen AM, Vera JF, Dotti G, Gee AP, Brenner MK, Myers DG, Rooney CM. Early transduction produces highly functional chimeric antigen receptor-modified virus-specific T-cells with central memory markers: a Production Assistant for Cell Therapy (PACT) translational application. J Immunother Cancer. 2015 Feb 18;3:5. doi: 10.1186/s40425-015-0049-1. eCollection 2015. PMID 25734008
- [Derived] Cruz CR, Micklethwaite KP, Savoldo B, Ramos CA, Lam S, Ku S, Diouf O, Liu E, Barrett AJ, Ito S, Shpall EJ, Krance RA, Kamble RT, Carrum G, Hosing CM, Gee AP, Mei Z, Grilley BJ, Heslop HE, Rooney CM, Brenner MK, Bollard CM, Dotti G. Infusion of donor-derived CD19-redirected virus-specific T cells for B-cell malignancies relapsed after allogeneic stem cell transplant: a phase 1 study. Blood. 2013 Oct 24;122(17):2965-73. doi: 10.1182/blood-2013-06-506741. Epub 2013 Sep 12. PMID 24030379